CLINICAL TRIAL: NCT03102281
Title: Gastrointestinal Microbiomes in Patients of Recurrent Common Bile Duct Stones After Endoscopic Sphincterotomy（EST）
Brief Title: Microbiomes in Patients of Recurrent Common Bile Duct Stones
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: BDS-CN-1702
Record Dates: First submitted 2017-03-08; First posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Cholelithiasis; Choledocholithiasis
MeSH Terms: conditions — Cholelithiasis; Choledocholithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- recurrent group: Patients who had recurrent common bile duct stones.
- control group: Patients who had not recurrent common bile duct stones.

SUMMARY:
Bile duct stones is a common biliary tract disease, which is characterized by high morbidity and frequent recurrence. Endoscopic retrograde cholangiopancreatography (ERCP) is an effective therapy for common bile duct stones, and endoscopic sphincterotomy (EST) which associated with recurrent cholangiolithiasis often carried out on difficult intubation or extracting stones, probably due to enhanced reflux of intestinal contents that changes the microenvironment. Patients with cholangiolithiasis were consecutively recruited and their bile was collected intra-operatively for high-throughput experiments. Pyrosequencing of 16S ribosomal RNA gene was performed to characterize the microbiota in the bile and other body fluids. A liquid chromatography mass spectrometry-based method was used to profile bile composition. Clinical manifestation, microbiome, and bile composition were compared between patients with or without recurrent of bile duct stones. The aim of our study was to identify the impact of microbiomes on the recurrent of bile duct stones after ERCP+EST therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recurrent common bile duct stones.
2. No antibiotics or probiotics are used for nearly three months.
3. In addition to common bile duct stones, possibly without other digestive diseases.

Exclusion Criteria:

1. Significant neurological or psychiatric disorders (psychotic disorders, dementia or seizures) that would prohibit the understanding and giving of informed consent.
2. Pregnant or lactating females.
3. Active Hepatitis B or C or history of an HIV infection.
4. Active uncontrolled infection.
5. Billroth II or roux-en Y gastrointestinal alteration people.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be adults with recurrent common bile duct stones.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes of Bacteria in Body Fluid | 3 years
  measure the changes of Bacteria in Body Fluid

SECONDARY OUTCOMES:
Stone diameter | 3 years
  measure the stone diameter
EST size | 3 years
  measure the EST size
Stone type | 3 years
  test the stone type
Bile acid composition(Mass spectrometry or Chromatography) | 3 years
  measure the bile acid composition with Mass spectrometry or Chromatography

CONTACTS AND LOCATIONS:
Overall Officials: Miao Lin, Study Principal Investigator, Principal Investigator — Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No